CLINICAL TRIAL: NCT01486303
Title: Efficacy and Safety of Facial Cosmetic Acupuncture on Skin Rejuvenation
Brief Title: Facial Cosmetic Acupuncture on Skin Rejuvenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyunghee University (Other)
Responsible Party: Principal Investigator, Inhwa Choi, Chief of Department of Oriental Dermatology, Kyunghee University Hospital at Gangdong, Kyunghee University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB2011-007
Record Dates: First submitted 2011-11-14; First posted 2011-12-06 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Skin Aging; Skin Wrinklings
Keywords: Facial Cosmetic acupuncture; Skin Rejuvenation; Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Facial Cosmetic Acupuncture (Experimental): 28 Patients with grade III to IV wrinkling on the face, according to the Glogau classification system, were treated with Facial Cosmetic Acupuncture.
  Interventions: Procedure: Facial Cosmetic Acupuncture

INTERVENTIONS:
Procedure: Facial Cosmetic Acupuncture — Patients received five treatment sessions during 3 weeks. Facial cosmetic acupuncture was applied at muscles and acupoints on the face, head and neck

SUMMARY:
Facial Cosmetic Acupuncture technique includes wrinkles, acupoints and muscle points on the face, head and neck. This study is designed to determine the efficacy and safety of Facial Cosmetic Acupuncture on skin rejuvenation.

ELIGIBILITY:
Inclusion Criteria:

* Patient age of 40 to 59 years
* Glogau photoaging scale III-IV

Exclusion Criteria:

* Who had undergone any dermabrasion, deep skin peels, laser resurfacing (ablative or non-ablative), botulinum toxin or filler injection, topical steroid within 6 months prior to study entry
* Patient with obvious skin disease
* Patient with a history of chronic skin disease
* Keloidal or hypertrophic scar tendency
* Pregnant or lactating patients

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Criteria for evaluating Moire's topography | At 3 weeks (post treatment)
  The investigators generated a contour line on the face using Moire's system, and then took a picture with a digital camera Ixus750 (Canon, Tokyo, Japan). Three independent evaluators will read the contour lines near the cheek and the perioral region in the printed digital image and grade images base on the Criteria for evaluating Moire's topography (Skin Research and Technology 2007;13:280-284). The average values from three evaluators will be used in subsequent calculations.

SECONDARY OUTCOMES:
Glogau classification system | At 3 weeks (post treatment)
One-click Automatic Full face Analysis system | At 3 weeks (post treatment)
  Improvement of Pore, Sebum, wrinkle, pigment, moisture, elasticity, skin temperature based on automatic analysis by Scanner and Multi-Sensor of One-click Automatic Full face Analysis system. Outcomes will be graded from 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hwa Choi, KMD,PhD, Study Chair — Department of Oriental Dermatology, College of Oriental Medicine, Kyung Hee University; Younghee Yun, KMD,Master, Principal Investigator — Department of Oriental Dermatology, College of Oriental Medicine, Kyung Hee University
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

REFERENCES:
- See also: Related Info — http://www.khnmc.or.kr